CLINICAL TRIAL: NCT06414603
Title: A Comparative Effectiveness Study in Heart Transplant Patients of Rejection Surveillance With Cell-free DNA Versus Endomyocardial Biopsy (ACES-EMB)
Brief Title: A Comparative Effectiveness Study in Heart Transplant Patients of Rejection Surveillance With Cell-free DNA Versus Endomyocardial Biopsy
Acronym: ACES-EMB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Natera, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-069-TRP
Record Dates: First submitted 2024-05-02; First posted 2024-05-16 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-08

CONDITIONS: Heart Transplant Failure and Rejection
Keywords: Heart Transplant
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prospera Surveillance Cohort (Experimental): Subjects are required to undergo Prospera testing at times corresponding to the institution's graft surveillance schedule. Prospera test results will be provided to the clinical team. Prospera cfDNA level < 0.15% will be interpreted as low risk for acute rejection (AR). Prospera cfDNA ≥ 0.15% will be interpreted as increased risk for AR and may be followed by EMB to rule out AR at the discretion of the treating clinicians. All other standard of care modalities for assessing AR can be used at the discretion of the treating clinicians at any time throughout the study.
  As per standard of care, in subjects with clinical signs or symptoms of rejection, a for cause EMB can be done per the clinical team's discretion at any time during the study.
  Interventions: Diagnostic Test: The Prospera™ Test
- Endomyocardial Biopsy Surveillance Cohort (No Intervention): Subjects will undergo surveillance EMB per the institution's standard clinical care. Biopsy interpretation will be per the institutional pathologist using international guidelines for grading of acute cellular or antibody-mediated rejection.
  Subjects will also have Prospera testing performed at the time of surveillance EMB for the purpose of measuring concordance between dd-cfDNA surveillance testing and surveillance EMB; Prospera results will not be returned to investigators for subjects in the EMB surveillance group.

INTERVENTIONS:
Diagnostic Test: The Prospera™ Test — The Prospera™ test is a non-invasive test intended to detect and quantify the fraction of donor-derived cell-free DNA (dd-cfDNA) to supplement management and surveillance of allograft rejection in patients who have undergone organ transplantation. It employs Next Generation Sequencing (NGS), which is performed on cell-free DNA (cfDNA) that is extracted from the patient's plasma to discriminate between the patient's DNA and the solid organ-allograft DNA.
  In study 23-069-TRP, the Prospera test is indicated for heart allograft rejection surveillance in lieu of surveillance endomyocardial biopsy. Prospera results should be considered together with clinical evaluations and other diagnostic testing or imaging results. Prospera will be run as a centralized laboratory developed test that is developed and validated under Design Controls. The test will be run within Natera's CLIA-certified and CAP-accredited laboratory.
  Arms: Prospera Surveillance Cohort

SUMMARY:
This is an open label Comparative Effectiveness Research (CER) study in which patients will be randomized at the site level to Prospera surveillance or EMB surveillance in a 2:1 ratio (Prospera to EMB) at each site.

Subjects will be enrolled into the study while under evaluation for heart transplantation or on the transplant waiting list prior to heart transplantation. All subjects will follow the center's standard of care surveillance schedule from transplant through 4 weeks post-transplantation. EMB during this phase is expected to occur roughly weekly or bi-weekly.

Study group assignment will take place at randomization. Subjects will be randomized 30 days (± 10 days) post-transplant to Prospera surveillance versus EMB surveillance in a 2:1 ratio. Rejection surveillance (Prospera Group and EMB Group) will be performed at times corresponding to the institutional standard of care schedule for rejection surveillance.

DETAILED DESCRIPTION:
All subjects will undergo standard of care assessments for rejection monitoring in addition to Prospera testing and/or EMB in accordance with each site's clinical care protocols and at the discretion of the treating clinician. Quality of life questionnaires will be completed at week 4, month 6 and month 12 post-transplant.

Study Group: Prospera (dd-cfDNA) Surveillance Group Subjects are required to undergo Prospera testing at times corresponding to the institution's graft surveillance schedule. Prospera test results will be provided to the clinical team. Prospera cfDNA level < 0.15% will be interpreted as low risk for acute rejection (AR). Prospera cfDNA ≥ 0.15% will be interpreted as increased risk for AR and may be followed by EMB to rule out AR at the discretion of the treating clinicians. All other standard of care modalities for assessing AR can be used at the discretion of the treating clinicians at any time throughout the study. As per standard of care, in subjects with clinical signs or symptoms of rejection, a for cause EMB can be done per the clinical team's discretion at any time during the study.

Control Group: EMB Surveillance Group Subjects will undergo surveillance EMB per the institution's standard clinical care. Biopsy interpretation will be per the institutional pathologist using international guidelines for grading of acute cellular or antibody-mediated rejection. Subjects will also have Prospera testing performed at the time of surveillance EMB for the purpose of measuring concordance between dd-cfDNA surveillance testing and surveillance EMB; Prospera results will not be returned to investigators for subjects in the EMB surveillance group.

Subjects in both the Prospera and EMB Surveillance Groups will have Prospera blood draws performed at the time of any for cause EMB. Results of Prospera testing performed in conjunction with for cause EMB will not be returned to investigators or subjects.

Blood samples for exploratory mechanistic endpoints (miRNA) will be obtained at the time of each Prospera or EMB surveillance visit and at the time of any for cause EMB.

The study period will be during the first 12 months post-transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older at the time of signing informed consent.
2. Undergoing transplant evaluation or currently on the heart transplant waiting list and expected to receive a heart transplant.
3. Able to read, understand and provide written informed consent. If the patient is unable to sign informed consent, a legally authorized representative (LAR) can consent on behalf of the patient.
4. Able and willing to comply with the study visit schedule, study procedures and study requirements.

Exclusion Criteria:

1. Concurrent multiple solid organ or tissue transplants.
2. Prior history of any organ or cellular transplantation.
3. Planned use of other commercially available or investigational cfDNA or gene expression profile assays for rejection surveillance.
4. Pregnant.
5. Hemodynamically unstable or other serious medical condition that may adversely affect the subject's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Primary Clinical Endpoint | 12 months
  Incidence of the composite endpoint defined as the first occurrence of treated rejection with graft dysfunction*, treated rejection without graft dysfunction, graft dysfunction, retransplantation, and/or death.
  Clinical endpoints are defined as follows:
  1. Rejection: ISHLT ACR Grade ≥ 2R or AMR Grade ≥ pAMR1
  2. Graft dysfunction: LVEF decline ≥ 10% from baseline and < 50% absolute LVEF by echocardiography
  3. Retransplantation: being listed for re-transplant or being re-transplanted
     * Treated rejection with graft dysfunction and/or graft dysfunction requiring treatment with pulse dose steroids, monoclonal antibodies, plasmapheresis, and/or intravenous immunoglobulin (IVIg).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Olymbios, MD, Study Director — Natera, Inc.; Josef Stehlik, MD, Study Chair — University of Utah; Palak Shah, MD, Study Chair — Inova Schar Heart and Vascular
Locations (11):
- United States (11):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - University of Colorado, Aurora, Colorado
  - Mayo Clinic, Jacksonville, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Duke University, Durham, North Carolina
  - University of Texas, Southwestern Medical Center, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - Inova Schar Heart and Vascular Institute, Falls Church, Virginia

REFERENCES:
- [Derived] Kim H, Cusi V, McLenon M, Rodriguez JBC, Bui QM, Chak J, Urey MA, Cole J, Fielding-Miller R, Kim PJ. Perspectives of Heart Transplant Patients and Providers on Acute Rejection Surveillance: A Mixed-Methods Study. Clin Transplant. 2026 Jan;40(1):e70438. doi: 10.1111/ctr.70438. PMID 41492943